CLINICAL TRIAL: NCT06339411
Title: Examining the Efficacy of Cerebrolysin-Augmented Extended Time Window Thrombectomy in Acute Ischemic Stroke: An In-depth Study of Blood-brain Barrier Biomarkers and Imaging Indicators
Brief Title: Exploring Cerebrolysin in Late Thrombectomy for Stroke: Blood-brain Barrier Biomarkers and Imaging Insights
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202302239A3
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — cerebrolysin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended Thrombectomy with Cerebrolysin (Experimental): Cerebrolysin 30milliliter/quaque die(QD) for 10~14days intravenous drip (IVD)
  Interventions: Drug: Cerebrolysin
- Extended Thrombectomy without Cerebrolysin (No Intervention): No cerebrolysin

INTERVENTIONS:
Drug: Cerebrolysin — Cerebrolysin post-mechanical thrombectomy, initiated within 24 hours of stroke onset and continued for 14 days. The study assessed neurological, neuropsychological, and biomarker outcomes at multiple time points post-stroke to evaluate the effects of Cerebrolysin on recovery.
  Arms: Extended Thrombectomy with Cerebrolysin

SUMMARY:
Background:

Stroke is a leading cause of mortality and disability globally, with acute ischemic strokes(AIS) due to Large Vessel Occlusion (LVO) presenting significant treatment challenges. Mechanical thrombectomy (MT) has emerged as an effective intervention for AIS within an 8-hour window from symptom onset. However, the potential to extend this window up to 24 hours for select patients could revolutionize outcomes for those arriving late at comprehensive stroke centers. This study investigates the efficacy and safety of Cerebrolysin as an adjunct therapy to MT in extended time window and improving patient recovery.

Methods:

We conducted a multi-center, prospective, randomized study within the Chang Gung Memorial Hospital system in Taiwan, targeting 100 AIS patients eligible for MT beyond the traditional 8-hour window. Participants were randomized to receive either standard care or Cerebrolysin post-MT, initiated within 24 hours of stroke onset and continued for 14 days. The study assessed neurological, neuropsychological, and biomarker outcomes at multiple time points post-stroke to evaluate the effects of Cerebrolysin on recovery.

Results:

The primary outcome will measure the proportion of patients achieving favorable functional outcomes (modified Rankin Scale 0-2) at 90 days. Secondary outcomes include the impact of Cerebrolysin on secondary hemorrhagic transformation, brain edema, mortality rates, and quality of life. The study aims to provide comprehensive data on the benefits of adding Cerebrolysin to the standard post-MT care, focusing on its potential to protect against reperfusion injuries and maintain blood-brain barrier integrity.

Conclusion:

By evaluating the role of Cerebrolysin in conjunction with MT, this study aims to extend the therapeutic window for AIS treatment, offering hope for improved outcomes for patients who would otherwise be ineligible for current reperfusion therapies. The findings may pave the way for new guidelines in stroke management, emphasizing the importance of integrated care approaches in enhancing patient recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients capable of initiating endovascular therapy between 8-24 hours after the time they were last known to be well.
* Age above 18 years.
* NIHSS (National Institutes of Health Stroke Scale) score of ≥6, indicating moderate to severe stroke.
* Presence of likely salvageable ischemic brain tissue, as determined by CT (Computed Tomography) with ASPECTs (Alberta Stroke Program Early CT Score) ≥3.
* Occlusion of the proximal MCA-M1 (middle cerebral artery - M1 segment) or ICA (internal carotid artery) detected on CT angiography.
* Infarct volume <70 ml on Perfusion CT.
* Ischemic tissue showing an infarct volume ratio ≥1.8 on Perfusion CT.
* Absolute volume of potentially reversible ischemia (penumbra) ≥15 ml.
* Minimal pre-existing disability, with a Modified Rankin Scale (mRS) score of 0-2

Exclusion Criteria:

* Pregnancy
* Pre-existing terminal or debilitating illness
* Seizure activity preventing accurate determination of NIHSS score
* Abnormal blood glucose levels, with values below 50mg/dl or above 400mg/dl
* Platelet count <50,000 or International Normalized Ratio (INR) >3, indicating abnormal blood clotting parameters
* Neuroimaging findings indicating unsuitability for the procedure, such as ASPECTS score <3 on non-contrast CT, presence of intracranial tumor, acute intracranial hemorrhage, or occlusions in multiple vascular territories.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Functional Recovery and Complication Rates Post-Thrombectomy | mRS at 90 days and 12 months; NIHSS at 0, 1, and 7 days; mortality and Barthel Index at 90 days and 12 months post-stroke.
  This study will assess functional recovery primarily through the proportion of subjects achieving a favorable outcome as defined by an mRS score of 0-2. Secondary measures of efficacy will include changes in NIHSS scores at acute (day 0), subacute (day 1), and early convalescent (day 7) phases post-stroke. The incidence of complications such as secondary intracranial hemorrhage (ICH) or hemorrhage transformation (HT), as well as brain edema with midline shift, will be monitored. Mortality rates and functional independence, measured by the Barthel Index, will be evaluated to provide a comprehensive assessment of patient recovery and treatment impact.

SECONDARY OUTCOMES:
Imaging and High cortical Functional Assessment Endpoints | Imaging endpoints will be quantified at 30 days (1 month) and at 90 days (3 months) post-stroke. For functional and mood assessments within the Cerebrolysin group, evaluations will be precisely scheduled at 30 days post-stroke to establish early recovery
  Secondary outcomes will include imaging endpoints to measure the impact of Cerebrolysin on cerebral tissue preservation, specifically evaluating final infarct volume, infarct growth, and penumbral salvage. Functional assessments will track changes in language function using the 15-item Boston Naming Test, global cognitive function via the Montreal Cognitive Assessment, and mood disturbances with the Hamilton Depression Rating Scale. These assessments will collectively inform on the neuroprotective effects of Cerebrolysin.

IPD SHARING:
Plan to Share IPD: No